CLINICAL TRIAL: NCT00028730
Title: Phase II Trial of T-Cell Depleted Hematopoietic Stem Cell Transplants (SBA-E-BM) From HLA Compatible Related or Unrelated Donors After a Myeloablative Preparative Regimen of Hyperfractionated TBI, Thiotepa and Cyclophosphamide (TBI/Thio/cy) for Treatment of Patients Less Than or Equal to 18 Years With Lymphohematopoietic Disorders
Brief Title: Total-Body Irradiation and Chemotherapy Followed By Donor Bone Marrow Transplant in Treating Young Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-105; P30CA008748 (NIH); P01CA033049 (NIH); P01CA023766 (NIH); MSKCC-01105; NCI-H01-0083
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: recurrent childhood lymphoblastic lymphoma; chronic phase chronic myelogenous leukemia; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Chronic-Phase; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; Filgrastim; Cyclophosphamide; fludarabine phosphate; Thiotepa; Radiotherapy

ARMS (1):
- Pts < than or = 18 years with lymphohematopoietic disorders (Experimental): This is a phase II, single-center study to evaluate a cytoreductive regimen of hyperfractionated TBI, thiotepa and cyclophosphamide (HFTBI/thio/cy) followed by infusions of SBA-E- T-cell depleted marrow in pediatric leukemia recipients of either HLA-identical or HLA-1Ag non-identical related or unrelated donors.
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: thiotepa; Procedure: allogeneic bone marrow transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving chemotherapy and total body irradiation before a donor bone marrow transplant helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin and removing the T cells from the donor cells before transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well total-body irradiation and chemotherapy followed by T-cell depleted donor bone marrow transplant works in treating young patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of hyperfractionated total body irradiation, thiotepa, and cyclophosphamide followed by T-cell-depleted allogeneic bone marrow transplantation in children with acute myeloid leukemia, acute lymphoblastic leukemia, chronic myelogenous leukemia, non-Hodgkin's lymphoma, or myelodysplastic syndromes.
* Correlate the progenitor cell dose and dose of clonable T cells with the incidence and quality of engraftment, extent of chimerism, incidence and severity of acute and chronic graft-versus-host disease, characteristics of hematopoietic and immunologic reconstitution, and overall and disease-free survival at 2 years in patients treated with this regimen.

OUTLINE: Patients undergo total body irradiation three times daily on days -9 to -7 and twice on day -6. Patients receive thiotepa IV over 4 hours on days -5 and -4 and cyclophosphamide IV over 30 minutes on days -3 and -2. Patients who cannot receive cyclophosphamide, due to prior hemorrhagic cystitis or exposure to high-dose cyclophosphamide or ifosfamide, receive fludarabine IV over 30 minutes on days -5 to -1. Patients planning to receive family member HLA-mismatched or unrelated bone marrow transplantation receive horse anti-thymocyte globulin IV once daily on days -5 and -4. Patients undergo allogeneic T-cell-depleted bone marrow transplantation on day 0. Patients receive filgrastim (G-CSF) IV every 12 hours beginning on day 7 and continuing until blood counts recover.

Patients are followed every 2-4 weeks for the first 100 days post-transplantation, every 6 weeks for 6 months, every 3 months for 1 year, and then every 3-6 months until 2 years post-transplantation.

PROJECTED ACCRUAL: A total of 50 patients (25 with HLA 6/6 antigen-matched related donors and 25 with HLA 5/6 antigen-matched related donors or HLA 5/6 or 6/6 antigen-matched unrelated donors) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically confirmed good-risk acute myeloid leukemia (AML) in first remission with an HLA-compatible related donor

    * Ineligible for unrelated bone marrow transplantation unless failed first-line induction chemotherapy or have molecular evidence of disease at time of transplantation
  * Histologically confirmed high-risk AML in first remission

    * High risk defined by cytogenetics, biphenotypic and undifferentiated leukemia phenotype, secondary AML, or AML after myelodysplastic syndromes (MDS)
    * Eligible for related or unrelated donor transplantation
  * Histologically confirmed acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LL) in first remission with high risk for relapse or in second or third remission

    * High risk for relapse defined by hypodiploidy, pseudodiploidy with translocations t(9;22) or infant t(4;11), or failure to achieve remission after four weeks of induction therapy
    * Eligible for related or unrelated donor transplantation
  * Histologically confirmed chronic myelogenous leukemia (CML) in at least first chronic phase or acceleration with an HLA-compatible related donor
  * Histologically confirmed CML in first chronic phase if failed conventional therapy or in at least second chronic phase or acceleration with an HLA-compatible unrelated donor
  * Histologically confirmed non-Hodgkin's lymphoma beyond first complete remission or primary induction failure and tumors that are chemosensitive defined as at least 50% reduction in mass size

    * Eligible for related or unrelated donor transplantation
  * Histologically confirmed MDS with intermediate or high-risk disease defined by International Prognostic Scoring System and paroxysmal nocturnal hematuria

    * Eligible for related or unrelated donor transplantation
* Treatment-related MDS or leukemia allowed if primary malignancy (e.g., neuroblastoma or Ewing's sarcoma) at low risk of recurrence
* No AML, ALL, or LL in relapse or greater than third remission
* No CML in blast crisis defined as more than 30% blasts plus promyelocytes
* No active CNS involvement
* History of leukemia cutis allowed
* HLA compatible donor available

  * 5/6 or 6/6 HLA antigen matched related or unrelated

PATIENT CHARACTERISTICS:

Age:

* 18 and under

Performance status:

* Karnofsky 70-100% OR
* Lansky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN (unless liver involvement is present)

Renal:

* Creatinine normal OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* LVEF at least 50% at rest (if less than 50% at rest, must increase with exercise)

Pulmonary:

* Asymptomatic with no prior risk features OR
* DLCO greater than 40% predicted (corrected for hemoglobin) if symptomatic

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV I/II negative
* No uncontrolled viral, bacterial, or fungal infection
* No known hypersensitivity to bovine proteins

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characterisitics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy that would preclude total body irradiation dose

Surgery:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2001-08; Primary Completion 2006-07 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Minimal transplantation related mortality | 2 years
High disease-free survival at 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Kernan, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States